CLINICAL TRIAL: NCT01178931
Title: Oral Dydrogesterone Versus Vaginal Progesterone Gel in the Luteal Phase Support: Randomized Controlled Trial
Brief Title: Dydrogesterone Versus Intravaginal Progesterone in the Luteal Phase Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Vlatka Tomic, MD, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KBSM-0010
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Luteal Phase Defect
Keywords: IVF; luteal phase support; oral progesterone; vaginal progesterone; pregnancy rate; safety; tolerability
MeSH Terms: interventions — Dydrogesterone; Crinone; Gels

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral dydrogesterone (Active Comparator): Study group receiving 2x10mg of oral dydrogesterone until a pregnancy test or in the case of pregnancy until 10 week.
  Interventions: Drug: Oral dydrogesterone
- Crinone 8% vaginal gel (Active Comparator): Control group is receiving vaginal gel, 1x90mg, until a pregnancy test or in the case of pregnancy until 10 week.
  Interventions: Drug: Crinone 8% gel

INTERVENTIONS:
Drug: Oral dydrogesterone — oral-2x10mg
  Other Names: Duphastone (Solvay Pharmaceuticals)
  Arms: Oral dydrogesterone
Drug: Crinone 8% gel — vaginal-1x90mg
  Other Names: Crinone 8% gel (Fleet Laboratories Ltd., Watford, UK)
  Arms: Crinone 8% vaginal gel

SUMMARY:
The purpose of this study is to compare efficacy and tolerability of the dydrogesterone and the vaginal progesterone, used for luteal phase support.

(Initial start date was January 2009 but not for patients' recruitment only for paper work, documents, team organization, statistical pre-work actions and to gain the official approval of Institutional Review Board. The recruitment started in October 2010 and continued until October 2013.)

DETAILED DESCRIPTION:
The use of gonadotropin-releasing hormone (GnRH) agonists in the ovarian stimulation, which prevents a premature surge of luteal hormone (LH), ultimately leads to suppression of the pituitary gland and high levels of estrogen observed during induced cycles result in inhibiting effect on the implantation of human embryos.

The luteal support in in-vitro-fertilization (IVF) cycles can be prolonged using human chorion gonadotropin(hCG) and/or progesterone.

Since it has been noted that the use of hCG was related with higher risks of the onset of ovarian hyperstimulation syndrome (OHSS), progesterone is nowadays a product of choice in luteal support.

Currently vaginal progesterone is widely used, since the classic oral progesterone results in low bioavailability and lower pregnancy rate and the intramuscular progesterone (IM-P) daily injections are painful and may cause abscesses, inflammatory reactions and local soreness.

However, standard protocol for luteal phase support has not been established (i.e. optimal dosage, route or duration).

Dydrogesterone is a retroprogesterone with good oral bioavailability. Oral administration is clear advantage, due to expected higher patient compliance and better tolerability than currently used vaginal or IM-P.

We hypothesize that dydrogesterone has the same efficacy as vaginal progesterone but better tolerability due to less side effects.

ELIGIBILITY:
Inclusion Criteria:

* routine ovulation induction protocol with GnRH agonist
* less than three prior IVF cycles
* at least three aspirated oocytes
* BMI <35 kg/m2
* age <45 years

Exclusion Criteria:

* history of dysfunctional uterine bleeding
* acute urogenital disease
* recurrent miscarriage
* previous allergic reactions to a progesterone products

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 853 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks
  Ongoing pregnancy rate is defined by the presence of gestational sac(s) with viable fetal heart beats at 12 weeks' gestation by transvaginal ultrasound.

SECONDARY OUTCOMES:
Number of participants with adverse events | 10 weeks
  The side effects included the occurrence of headache, somnolence, nausea, abdominal pain, bloating, dizziness, headache, breast fullness, perineal irritation, vaginal discharge and bleeding, interference with coitus.
Satisfaction | 10 weeks
  Satisfaction score is determinate on the 5-point level scale with 1 being "absolutely satisfied" and 5 being "absolutely dissatisfied" and tolerability by yes and now answers regarding side effects that the supplements could cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jozo Tomic, M.D., Principal Investigator — Department of Human Reproduction, University Hospital Center Sisters of Mercy; Vlatka Tomic, M.D., Study Chair — Department of Human Reproduction, University Hospital Center Sisters of Mercy
Locations (1):
- University Hospital Center Sisters of Mercy, Zagreb, Croatia

REFERENCES:
- [Derived] Tomic V, Tomic J, Klaic DZ, Kasum M, Kuna K. Oral dydrogesterone versus vaginal progesterone gel in the luteal phase support: randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2015 Mar;186:49-53. doi: 10.1016/j.ejogrb.2014.11.002. Epub 2014 Nov 20. PMID 25622239